CLINICAL TRIAL: NCT05582889
Title: Improving Physical Functioning in Older Cancer Survivors Through Light-Intensity Physical Activity
Brief Title: Move For Your Health for Older Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: UNM HSC 17-335; K07CA215937 (NIH)
Record Dates: First submitted 2022-09-27; First posted 2022-10-17 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Cancer Survivors
Keywords: cancer survivor; physical activity; sedentary behavior; cancer survivorship; rural; older; Hispanic; physical function; physical performance; quality of life; home-based; distance-based
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Immediate Fitbit Intervention (Experimental): Participants randomized to this arm receive the 12-week Fitbit intervention; participants then crossover and are observed (no health coaching) for an additional 12-weeks. The Fitbit intervention includes a Fitbit activity tracker, the free Fitbit smartphone app, and 6 Health Coaching calls.
  Interventions: Behavioral: Fitbit Intervention
- Comparator: Delayed Fitbit Intervention (Active Comparator): Wait-listed; participants maintain their usual physical activity for 12-weeks; participants then crossover and receive the full 12-week Fitbit intervention.
  Interventions: Behavioral: Fitbit Intervention

INTERVENTIONS:
Behavioral: Fitbit Intervention — Participants receive a Fitbit activity tracker and the free Fitbit smartphone app. A trained health coach provides technical support to set up and use the Fitbit and app. The health coach also provides motivational counseling to help participants to gradually increase the number of steps per day during the 12-weeks.

SUMMARY:
The Move for Your Health (MY Health) Pilot Study is a 12-week study for older cancer survivors to promote light physical activity. The home-based study (no travel required) will test whether a Fitbit activity tracker and health coaching can help cancer survivors be more active throughout the day.

DETAILED DESCRIPTION:
The objective is to examine the feasibility and acceptability of a home-based lifestyle activity intervention to promote light-intensity activity using a whole-of-day approach. Sixty-four older cancer survivors will be randomized to either a 12-week theory-based intervention or a waitlist control. The intervention uses a Fitbit activity tracker that pairs with a smartphone app to promote awareness and enable self-monitoring of both activity and inactivity. Motivational counseling will be used to individually tailor strategies to achieve goals. Data will be collected at baseline, post-intervention (week 13), and 3-months post-intervention (week 26).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed in New Mexico (NM) with a loco-regionally staged cancer, completed primary treatment (surgery, radiation, chemotherapy), and not currently being treated for a recurrence. Patients with metastatic cancer are eligible with physician approval.
* Mild-to-moderate physical functional impairment (raw score between 20 and 34 on the 8-item PROMIS Physical Function survey)
* Able to speak, read, & understand English or Spanish
* Participating in less than 120 minutes per week of moderate-intensity physical activity
* Living independently and capable of walking 3 blocks (approximately 1300 steps or 0.25 mile) without an assistive device (e.g., cane, walker) and without stopping to rest
* Own a smartphone or tablet *OR* be willing to use a study-provided smartphone capable of running the Fitbit app. Also, access to the internet or a Wi-Fi hotspot at least once per week is required. Smartphones and data plans will be provided to those individuals who are eligible but do not currently own a device capable of running the Fitbit app.
* Availability of a family member or friend to be present (for safety) during the remote assessment of physical performance tests
* Willingness to be randomized to either study arm and to wear activity trackers

Exclusion Criteria:

* Adults not able to consent
* Severe impairments (in seeing or hearing) or pre-existing medical limitations for engaging in daily light physical activity (e.g., severe orthopedic conditions, pending hip/knee replacement, dementia, oxygen dependent, chronic vertigo)
* Paid employment or volunteer position for greater than 20 hours per week (to avoid potential confounding by occupation activity/inactivity)
* Currently participating in a program (personal program, e.g., wearing an activity monitor, or structured program, e.g., another study) to decrease sedentary time or increase physical activity
* Planning to move out of New Mexico within the next year

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy K Blair, PhD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Blair CK, Brown-Glaberman U, Walters ST, Pestak C, Boyce T, Barriga L, Burgess E, Tawfik B, Killough C, Kinney AY, Demark-Wahnefried W, Meisner AL, Wiggins CL, Pankratz VS, Davis S. A Remotely Delivered Light-Intensity Physical Activity Intervention for Older Cancer Survivors: Protocol for a Feasibility Randomized Controlled Trial. JMIR Res Protoc. 2024 Dec 13;13:e59504. doi: 10.2196/59504. PMID 39671575

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Started | 32 | 32
Completed | 27 | 26
Not Completed | 5 | 6
Not completed — Health event | 3 | 2
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.6 (6.4) | 72.0 (5.0) | 72.8 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 8 | 10 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race-ethnicity: Hispanic | 10 | 10 | 20
  Race-ethnicity: non-Hispanic White | 20 | 20 | 40
  Race-ethnicity: Other | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Time to Accrual Goal
Description: The number of months to accrue the study sample. Accrual is part of assessing feasibility.
Time Frame: up to 1-year
Measure: Number; unit: months
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
months | 9 | 9

2. Primary Outcome: Study Participant Retention Rate
Description: The proportion of participants who complete the study out of the number randomized to one of two study arms. Retention is part of assessing feasibility.
Time Frame: 24-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
Participants | 27 | 26

3. Primary Outcome: Study Participant Adherence Rate
Description: The proportion of participants who complete all five health coaching calls and wear the Fitbit activity tracker at least 67 days (67 days = 80% x 12 weeks). Adherence is part of assessing feasibility.
Time Frame: 24-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
Participants | 29 | 26

4. Primary Outcome: Number of Adverse Events Attributable to the Study
Description: The number of adverse events attributable to or possibly attributable to the intervention will be tracked; defined as any condition that is life-threatening and results in overnight hospitalization or a physical or cardiac event serious enough to require medical attention. The number of adverse events is part of assessing feasibility.
Time Frame: 12-weeks
Measure: Number; unit: adverse events
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
adverse events | 0 | 0

5. Primary Outcome: Change in Self-reported Physical Function
Description: Self-reported physical function will be assessed using the PROMIS® Item Bank v2.0 - Physical Function - Short Form 8b. Raw scores range from 8 to 40, with higher scores indicative of better physical functioning.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | 0.03 (4.25) | 1.22 (3.77)

6. Secondary Outcome: Change in the Number of Chair Stands During the 30-second Chair Stand Test
Description: Physical performance will be objectively measured using the 30-second chair stand test, measured by the number of times a person comes to a full standing position from a chair in 30 seconds. Scores range from zero (cannot perform the test) to 30 or higher, with a higher number of chair stands representing stronger leg strength.
Time Frame: 12-weeks
Measure: Median (Inter-Quartile Range); unit: chair stands
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
chair stands | 1.0 [-1.0 to 2.0] | 0.5 [-0.5 to 1.0]

7. Secondary Outcome: Change in Balance Score During the 4-stage Balance Test.
Description: Physical performance will be objectively measured using the 4-stage balance test. The 4-stage balance test includes standing in each of four positions for up to 10 seconds: 1) feet side-by-side; 2) semi-tandem stand [one foot slightly behind but touching the other foot]; 3) tandem stand [one foot in front of the other; heel touching toe]; and 4) stand on one foot. Scores range from zero (participant refused, failed, or excluded from side-by-side test) to 5 (all four positions held for maximum time). Higher scores represent better balance.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | 0.0 (0.5) | 0.1 (0.5)

8. Secondary Outcome: Change in Number of Steps Per Day
Description: The activPAL accelerometer/inclinometer will be used to measure steps per day. Participants will be asked to wear the monitor for 7-days. Average daily steps will be calculated as the total steps divided by the number of days the monitor was worn.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 31 | 31
steps per day | 1168 (2285) | 69 (1495)

9. Secondary Outcome: Change in Objective Measures of Light-intensity Physical Activity
Description: The activPAL accelerometer/inclinometer will measure the daily minutes spent in light-intensity stepping. The average daily minutes of light-intensity stepping will be the total minutes divided by the number of days the activPAL monitor was worn. Light-intensity stepping is defined as stepping at a cadence between 75 and 99 steps per minute.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 31 | 31
minutes per day | 16.4 (30.7) | 0.0 (14.5)

10. Secondary Outcome: Change in Objective Measures of Moderate-intensity Physical Activity
Description: The activPAL accelerometer/inclinometer will measure the daily minutes spent in moderate-intensity stepping. The average daily minutes of moderate-intensity stepping will be the total minutes divided by the number of days the activPAL monitor was worn. Moderate-intensity stepping is defined as stepping at a cadence of at least 100 steps per minute.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 31 | 31
minutes per day | 8.7 (17.4) | -1.1 (7.0)

11. Secondary Outcome: Change in Objective Measures of Sedentary Activity
Description: The activPAL accelerometer/inclinometer will measure minutes spent in sedentary activities (not including sleep). The average daily minutes of sedentary time will be the total minutes divided by the number of days the activPAL monitor was worn.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 31 | 31
minutes per day | -24.6 (83.1) | 2.9 (57.4)

12. Secondary Outcome: Change in Self-reported Fatigue
Description: Self-reported fatigue will be assessed using the PROMIS® Item Bank v1.0 - Fatigue - Short Form 8a. Raw scores range from 8 to 40, with higher scores indicative of worse fatigue.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | -1.38 (5.76) | 1.09 (3.79)

13. Secondary Outcome: Change in Self-reported Pain
Description: Self-reported pain will be assessed using the PROMIS® Item Bank v1.0 - Pain Interference - Short Form 8a. Raw scores range from 8 to 40, with higher scores indicative of worse pain.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | 1.38 (7.38) | -0.56 (4.28)

14. Secondary Outcome: Change in Self-reported Sleep Disturbance
Description: Self-reported sleep disturbance will be assessed using the PROMIS® Item Bank v1.0 - Sleep Disturbance - Short Form 8b. Raw scores range from 8 to 40, with higher scores indicative of greater sleep disturbance.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | -0.78 (5.74) | 0.50 (4.59)

15. Secondary Outcome: Change in Self-reported Sleep Impairment
Description: Self-reported sleep impairment will be assessed using the PROMIS® Item Bank v1.0 - Sleep-Related Impairment - Short Form 8a. Raw scores range from 8 to 40, with higher scores indicative of greater sleep impairment.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | 0.81 (2.98) | 0.28 (4.88)

16. Secondary Outcome: Change in Self-reported Social Participation
Description: Self-reported ability to participate in social roles and activities will be assessed using the PROMIS® Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 8a. Raw scores range from 8 to 40, with higher scores indicative of greater social participation.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | 1.22 (6.93) | 0.06 (5.78)

17. Secondary Outcome: Change in Self-reported Anxiety
Description: Self-reported anxiety will be assessed using the PROMIS® Item Bank v1.0 - Emotional Distress - Anxiety - Short Form 8a. Raw scores range from 8 to 40, with higher scores indicative of greater anxiety.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | 0.91 (3.11) | -0.25 (4.47)

18. Secondary Outcome: Change in Self-reported Depression
Description: Self-reported depression will be assessed using the PROMIS® Item Bank v1.0 - Emotional Distress - Depression - Short Form 8a. Raw scores range from 8 to 40, with higher scores indicative of greater depression.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | 1.28 (4.17) | 0.03 (3.11)

19. Other Pre Specified Outcome: Change in Fall Risk
Description: Risk for falls will be assessed by the Falls Efficacy Scale International. Scores range from 16 to 64, with higher scores representing greater concern about falling.
Time Frame: 12-weeks
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | 0.0 [-2.0 to 1.0] | 0.0 [-2.0 to 2.0]

20. Other Pre Specified Outcome: Change in Fall Risk
Description: as for outcome 19
Time Frame: 24-weeks
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | 0.0 [-1.5 to 0.5] | 0.0 [-1.0 to 1.0]

21. Other Pre Specified Outcome: Change in Social Support for Physical Activity
Description: 4 items using a 5-point scale to measure support from family and friends while making changes to physical activity. Response items include never, once, sometimes, almost every day, and every day. Total scores range from 0 to 16; higher scores are indicative of greater social support for physical activity.
Time Frame: 12-weeks
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | 0.0 [-1.0 to 1.5] | 0.0 [-1.5 to 2.0]

22. Other Pre Specified Outcome: Change in Social Support for Physical Activity
Description: 4 items using a 5-point scale to measure support from family and friends while making changes to physical activity. Response items include never, once, sometimes, almost every day, and every day. Higher scores are indicative of greater social support for physical activity.
Time Frame: 24-weeks
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | 0.0 [-1.0 to 2.0] | 0.0 [-1.5 to 2.5]

23. Other Pre Specified Outcome: Change in Outcome Expectations
Description: Multidimensional Outcome Expectations for Exercise Scale includes 15 items to assess physical, social, and self-evaluative beliefs about the consequences of being physically active. Response items include strongly disagree, disagree, neutral, agree, and strongly agree. Scores range from 15 to 75, with higher scores indicative of higher levels of outcome expectations for exercise.
Time Frame: 12-weeks
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | 0.0 [-3.0 to 3.0] | -1.0 [-3.0 to 3.0]

24. Other Pre Specified Outcome: Change in Outcome Expectations
Description: as for outcome 23
Time Frame: 24-weeks
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | -1.0 [-5.0 to 2.0] | 0.0 [-4.0 to 4.0]

25. Other Pre Specified Outcome: Change in Motivation
Description: Behavioral Regulations in Exercise Questionnaire (BREQ-2) is a 19-item survey to assess autonomous motivation for exercise on a continuum from amotivation to intrinsic motivation. Mean scores range from 0 (not true for me) to 4 (very true for me) regarding motivation for exercise. Change in BREQ2 Relative Autonomy Index (RAI) is a single score derived from subscales. Subscales are weighted; RAI provides the degree to which a participant feels self-determined. Higher, positive scores indicate greater relative autonomy; whereas lower negative scores indicate more controlled regulation.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | 1.1 (4.2) | -0.4 (2.6)

26. Other Pre Specified Outcome: Change in Motivation
Description: Behavioral Regulations in Exercise Questionnaire (BREQ-2) is a 19-item survey to assess autonomous motivation for exercise on a continuum from amotivation to intrinsic motivation. Mean scores range from 0 (not true for me) to 4 (very true for me) regarding motivation for exercise. Behavioral Regulations in Exercise Questionnaire (BREQ-2) is a 19-item survey to assess autonomous motivation for exercise on a continuum from amotivation to intrinsic motivation. Mean scores range from 0 (not true for me) to 4 (very true for me) regarding motivation for exercise. Change in BREQ2 Relative Autonomy Index (RAI) is a single score derived from subscales. Subscales are weighted; RAI provides the degree to which a participant feels self-determined. Higher, positive scores indicate greater relative autonomy; whereas lower negative scores indicate more controlled regulation.
Time Frame: 24-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | -1.2 (4.3) | 1.6 (2.6)

27. Other Pre Specified Outcome: Perceived Autonomy Support
Description: Perceived Autonomy Support - Sport Climate Questionnaire (short form) includes 15 items to assess autonomy support of the health coach to characterize the quality of the social environment for influencing motivation to exercise. Mean individual scores range from 1 to 7, with higher scores indicating greater autonomy support from the health coach. Total score ranges from 7 (low autonomy) to 105 (high autonomy). Measured after the intervention for both groups; note: this survey was not administered prior to the intervention.
Time Frame: post-intervention (end of 12-week intervention)
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 26 | 26
points | 101.5 [96.0 to 105.0] | 99.0 [96.0 to 105.0]

28. Other Pre Specified Outcome: Change in Self-reported Physical Function
Description: as for outcome 5
Time Frame: 24-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | 1.31 (3.93) | 0.22 (3.89)

29. Other Pre Specified Outcome: Change in the Number of Chair Stands During the 30-second Chair Stand Test
Description: as for outcome 6
Time Frame: 24-weeks
Measure: Median (Inter-Quartile Range); unit: chair stands
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
chair stands | 0.0 [0.0 to 1.0] | 0.0 [0.0 to 1.0]

30. Other Pre Specified Outcome: Change in Balance Score During the 4-stage Balance Test.
Description: as for outcome 7
Time Frame: 24-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | 0.1 (0.5) | 0.0 (0.6)

31. Other Pre Specified Outcome: Change in Number of Steps Per Day
Description: as for outcome 8
Time Frame: 24-weeks
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 31 | 31
steps per day | 296 (1828) | 542 (2699)

32. Other Pre Specified Outcome: Change in Objective Measures of Light-intensity Physical Activity
Description: as for outcome 9
Time Frame: 24-weeks
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 31 | 31
minutes per day | 6.3 (24.4) | 9.8 (26.6)

33. Other Pre Specified Outcome: Change in Objective Measures of Moderate-intensity Physical Activity
Description: as for outcome 10
Time Frame: 24-weeks
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 31 | 31
minutes per day | 3.3 (11.6) | 5.2 (16.4)

34. Other Pre Specified Outcome: Change in Objective Measures of Sedentary Activity
Description: as for outcome 11
Time Frame: 24-weeks
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 31 | 31
minutes per day | -10.1 (66.5) | -4.4 (58.1)

35. Other Pre Specified Outcome: Change in Self-reported Fatigue
Description: as for outcome 12
Time Frame: 24-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | -0.31 (4.20) | -2.97 (6.31)

36. Other Pre Specified Outcome: Change in Self-reported Pain
Description: as for outcome 13
Time Frame: 24-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | 0.41 (6.63) | -0.91 (5.01)

37. Other Pre Specified Outcome: Change in Self-reported Sleep Disturbance
Description: as for outcome 14
Time Frame: 24-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | -0.78 (4.71) | -2.38 (4.51)

38. Other Pre Specified Outcome: Change in Self-reported Sleep Impairment
Description: as for outcome 15
Time Frame: 24-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | 0.22 (3.89) | -1.09 (4.00)

39. Other Pre Specified Outcome: Change in Self-reported Social Participation
Description: as for outcome 16
Time Frame: 24-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | -1.28 (5.59) | 1.00 (5.31)

40. Other Pre Specified Outcome: Change in Self-reported Anxiety
Description: as for outcome 17
Time Frame: 24-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | -0.75 (3.10) | -0.47 (3.93)

41. Other Pre Specified Outcome: Change in Self-reported Depression
Description: as for outcome 18
Time Frame: 24-weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
points | -1.94 (4.83) | 0.19 (2.97)

42. Primary Outcome: Number of Adverse Events Attributable to the Study
Description: as for outcome 4
Time Frame: 24-weeks
Measure: Number; unit: adverse events
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
Number analyzed (Participants) | 32 | 32
adverse events | 0 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Experimental: Immediate Fitbit Intervention | Comparator: Delayed Fitbit Intervention
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 1/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Immediate Fitbit Intervention (N=32) | Comparator: Delayed Fitbit Intervention (N=32)
Fall (General disorders) | 0 (0) | 1 (1) — The fall occurred among a participant in the waitlisted intervention during the delivery of the intervention (vs. the waitlisted period).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT05582889/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT05582889/ICF_001.pdf